CLINICAL TRIAL: NCT01490970
Title: Sarcoma Database at KFSH&RC.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: RAC# 2081-015; RAC# 2081-015
Record Dates: First submitted 2011-12-11; First posted 2011-12-13 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Sarcoma Database
Keywords: Sarcoma Database
MeSH Terms: interventions — Database Management Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Database — Database

SUMMARY:
Sarcoma Database

DETAILED DESCRIPTION:
Sarcoma Database

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed Sarcoma

Exclusion Criteria:

* Patients with diagnosis other than Sarcoma

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sarcoma Database
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2008-04; Primary Completion 2018-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: M Memon, M.D., Principal Investigator — KFSH & RC
Locations (1):
- Kfsh & Rc, Riyadh, Saudi Arabia